CLINICAL TRIAL: NCT03753867
Title: Retinoic Acid Effect on Cell Surface Molecules in Vivo
Brief Title: RA Effect on Cell Surface Molecules in Vivo
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was withdrawn.
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018 0639
Record Dates: First submitted 2018-10-01; First posted 2018-11-27 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Acitretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acitretin treatment (Experimental)
  Interventions: Drug: Acitretin

INTERVENTIONS:
Drug: Acitretin — Acitretin will be provided to participants in the formulation Soriatane. Soriatane doses are oral tablets taken daily by the participant. Participants will then receive 35mg of oral acitretin (Soriatane) daily for 8 weeks during the intervention phase. Participants will be asked to return two months after completion of the acitretin course for clinical follow-up and additional phlebotomy for laboratory testing.

SUMMARY:
This study will follow a group of healthy male participants for about 18 weeks to see the effect of taking Acitretin on their immune cells

DETAILED DESCRIPTION:
Retinoids have been shown in in vitro and ex vivo models to have the ability to reverse latency reactivating the HIV reservoir and the potential for selective eradication of HIV-harbouring cells. We feel that acitretin shows significant potential as a potential adjuvant to current ART regimens, however, there is a lack of data to demonstrate that treatment with acitretin at normal are able to induce molecular and transcription changes consistent with the above activities. In order to provide a scientific basis for retinoid therapy in HIV infection, a Phase I trial of acitretin in human subjects is proposed.

ELIGIBILITY:
Inclusion Criteria:

1. Male gender
2. Age 18 - 65
3. Able to provide informed consent
4. Willingness to participate in study treatment and follow-up
5. Willingness for serial phlebotomy and storage and future viro-immunological assays

Exclusion Criteria:

1. Female gender
2. Participants with a known hypersensitivity/allergy to the acitretin.
3. Participants who are actively participating in an experimental therapy study or who have received experimental therapy within the last 1 year.
4. Participants who are a poor medical risk because of other systemic diseases or active uncontrolled infections including HIV, Hepatitis B or C, and tuberculosis
5. Participants with impaired glucose tolerance including prediabetes or diabetes mellitus, dyslipidemia, or liver dysfunction
6. Previous or current history of mood disorder, psychosis, or suicidality
7. Participants currently receiving ongoing treatment with methotrexate, tetracyclines, or other retinoids

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-01-07 (Estimated); Primary Completion 2019-05-08 (Estimated); Study Completion 2019-05-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 5 months
  Safety of Acitretin use in healthy volunteers will be assessed using safety labs and C-SSRS

SECONDARY OUTCOMES:
Change in α4β7 expression on peripherally circulating CD4 T cells | Serial phlebotomy measured over 5 months
  Absolute change in α4β7 expression on peripherally circulating CD4 T cells measured using flow cytometry
Maximum Plasma Concentration [Cmax] | Trough concentrations measured serially over 2 months of active treatment
  Serum concentrations measured by HPLC
Change in RIG-1 expression, p300 expression, mTOR expression | Serial phlebotomy measured over 5 months
  Absolute change in RIG-1 expression by qRTPCR, and change in p300 expression by western blot, change in mTOR expression by qRTPCR and mTOR total/phosphorylated by western blot
Area Under the Curve [AUC]). | Trough concentrations measured serially over 2 months of active treatment
  Serum concentrations measured by HPLC

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B Angel, MD, FRCPC, Principal Investigator — Ottawa Hospital Research Institute

IPD SHARING:
Plan to Share IPD: Undecided